CLINICAL TRIAL: NCT03377114
Title: The Effect of Head Tilting on the Passing of Tracheal Tube Through Nasopharynx During Nasotracheal Intubation
Brief Title: Effect of Head Tilting During Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-2017-64
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Intubation;Difficult
Keywords: Nasotracheal intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutral (Active Comparator): When inserting a tracheal tube to oral cavity via nostril before use of laryngoscope in nasotracheal intubation, clinicians advance the tube with patient' head and neck in neutral position.
  Interventions: Procedure: Neutral
- Head tilting (Experimental): When inserting a tracheal tube to oral cavity via nostril before use of laryngoscope in nasotracheal intubation, clinicians advance the tube with patient' head in head-tilting position.
  Interventions: Procedure: Head tilting

INTERVENTIONS:
Procedure: Neutral — When inserting a tracheal tube to oral cavity via nostril before use of laryngoscope in nasotracheal intubation, clinicians advance the tube with patient' head and neck in neutral position.
  Arms: Neutral
Procedure: Head tilting — When inserting a tracheal tube to oral cavity via nostril before use of laryngoscope in nasotracheal intubation, clinicians advance the tube with patient' head in head-tilting position.
  Arms: Head tilting

SUMMARY:
The goal of this prospective randomized controlled study is to investigate the effect of head tilting on tracheal tube passing during nasotracheal intubation.

The question which the investigators are trying to answer is: If patient's neck is extented on inserting tracheal tube via nostril, will the E-tube be more easily to pass through nasopharynx to oropharynx without trapping?

DETAILED DESCRIPTION:
For nasotracheal intubation, clinicians do sometimes experience tube trapping at naso/oro-pharyngeal tissue. Application of force to overcome resistance can cause tissue injury leading to bleeding, which can disturb tracheal intubation.

The hypothesis of this study is that the method of 'head tilting' can help easy passing of tracheal tube at naso/oro-pharyngeal pathway without trapping in nasotracheal intubation. The purpose of the present study is to investigate the effect of 'head tilting' on the incidence of trapping of tracheal tube at naso/oro-pharynx when tracheal tube is being advanced into oropharynx via nostril during nasotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* The patients who need to nasotracheal intubation for surgery.

Exclusion Criteria:

* Who doesn't agree to enroll
* Who has a problem to head tilting position such as C-spine injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Tube trapping | During nasotracheal intubation
  When inserting a tracheal tube to oral cavity via nostril before use of laryngoscope in nasotracheal intubation, clinicians feel resistance in advancement.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Boramae Hospital, Seoul, South Korea

REFERENCES:
- [Background] Paul M, Dueck M, Kampe S, Petzke F, Ladra A. Intracranial placement of a nasotracheal tube after transnasal trans-sphenoidal surgery. Br J Anaesth. 2003 Oct;91(4):601-4. doi: 10.1093/bja/aeg203. PMID 14504169
- [Background] Bozdogan N, Sener M, Yavuz H, Yilmazer C, Turkoz A, Arslan G. Retropharyngeal submucosal dissection due to nasotracheal intubation. B-ENT. 2008;4(3):179-81. PMID 18949966
- [Background] Ersoy B, Gursoy T, Celebiler O, Umuroglu T. A complication of nasotracheal intubation after mandibular subcondylar fracture. J Craniofac Surg. 2011 Jul;22(4):1527-9. doi: 10.1097/SCS.0b013e31821d4e04. PMID 21778857
- [Derived] Kim H, Lee JM, Lee J, Hwang JY, Chang JE, No HJ, Won D, Row HS, Min SW. Effect of neck extension on the advancement of tracheal tubes from the nasal cavity to the oropharynx in nasotracheal intubation: a randomized controlled trial. BMC Anesthesiol. 2019 Aug 17;19(1):158. doi: 10.1186/s12871-019-0831-6. PMID 31421677